CLINICAL TRIAL: NCT02384031
Title: Quincke vs. Sprotte and Post-dural Puncture Headache - a Randomised Controlled Trial
Brief Title: Post-dural Puncture Headache - Needles and Biomarkers in CSF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: Imperial College London (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2011/1083/REK nord
Record Dates: First submitted 2015-02-27; First posted 2015-03-10 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Post-dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traumatic group (Active Comparator): Traumatic needle
  Interventions: Device: Traumatic needle
- Atraumatic group (Active Comparator): Atraumatic needle
  Interventions: Device: Atraumatic needle

INTERVENTIONS:
Device: Traumatic needle — Lumbar puncture is performed with a traumatic needle
  Other Names: Spinocan® (Quincke) 22Gx3.5"
  Arms: Traumatic group
Device: Atraumatic needle — Lumbar puncture is performed with an atraumatic needle
  Other Names: Pencan® (Sprotte) 22Gx3.5"
  Arms: Atraumatic group

SUMMARY:
Post-dural puncture headache (PDPH) is the most common complication following lumbar puncture (LP). The frequency varies widely depending on a number of factors, among which patient characteristics, case ascertainment, gauge and type of needle used are of significant importance. In 2001, Strupp et al. showed that over 12 % of 115 patients who were subjected to diagnostic lumbar puncture with a 22 gg (0.7 mm) atraumatic needle suffered post-dural puncture headache, while over 24 % of 115 who were given a lumbar puncture with a 22 gg traumatic needle suffered a headache. This finding provided the basis for an American recommendation to use a 22 gg atraumatic needle for diagnostic lumbar puncture. A later study with 58 patients has shown an even greater difference (36 % versus 3 % post-dural puncture headache) when an atraumatic needle is used. Despite these findings, European Neurologist continue to hold on to the cutting needle. Here the investigators propose a prospective randomized study design with double masking; neither patient nor evaluator of PDPH aware of the needle design used, and with an active ascertainment of the occurrence of PDPH in accordance with updated headache classification guidelines. The investigators also intend to investigate whether specific neuroinflammatory substances and metabolites (different outcome variables) in the cerebrospinal fluid (CSF) will affect the explanatory variable.

DETAILED DESCRIPTION:
Subjects are patients scheduled for a diagnostic LP as part of their routine clinical management at the department of Neurology, Nordland Hospital in Bodø, Norway. Selection is based on the inclusion and exclusion criteria listed beneath, independent of the primary clinical indication for the procedure.

Informed consenting patients will be randomised in two groups based on needle type. The traumatic group using Spinocan® (Quincke) 22Gx3.5" needle and atraumatic group using Pencan® (Sprotte) 22Gx3.5" needle. The randomisation process will be via an internet web-based application, provided by Norwegian university of science and Technology (http://www.ntnu.edu/dmf/akf/randomisering).

Subjects will undergo standard lumbar puncture, all in lateral recumbent position, the needle inserted, preferentially in level L3-4, perpendicular or parallel to the dural fibers, and CSF will be collected in accordance with the study protocol. Information about the LP, eventual complications, CSF volumes tapped and standard CSF-findings are noted.

Follow-up will be performed by investigators that are masked to the randomization. Patients will be interviewed over the telephone, alternatively in person if hospitalised, the first 1 and 7th day after the LP.Subjects that do develop PDPH will be treated in-line with established and standardized protocols at the department of Neurology, Nordland Hospital Trust, Bodø. Given that PDPH has a natural history of spontaneous resolution within 1-12 days, patients suffering from PDPH will be treated conservatively for the duration of the first 7 days after PDPH diagnosis. Conservative therapy, based on symptoms severity and patients' responsiveness, consist of the following: bed rest, caffeine, analgesics (paracetamol, NSAIDS), antiemetics and i.v. hydration. If the headache is severe and disabling and non-respondent after 7 days of conservative therapy, epidural blood patch will be administered. If a patient diagnosed with PDPH has a change in the pain character, or develops additional neurological manifestations, an urgent brain CT scan or MRI is indicated to exclude rarer potentially life-threatening intracranial complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at Department of Neurology, Nordland Hospital Trust in Bodø, scheduled for diagnostic LP

Exclusion Criteria:

1. Dementia
2. Non-compliance or coma
3. Local skin infections over proposed puncture site
4. Suspicion of raised intracranial pressure due to neurological or radiological findings
5. Bleeding diathesis (thrombocytopenia <50 x 109/L) or ongoing anticoagulant therapy
6. Major spinal column deformities
7. Procedural complications whereby needle type or size change is a requisite
8. Recent LP (< 7 days)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2012-02; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Post-dural puncture headache (PDPH) | At day 7 post LP

SECONDARY OUTCOMES:
Levels of neuropeptides in CSF | During lumbar puncture
Levels of metabolites in CSF | During lumbar puncture
Levels of inflammatory mediators in CSF | During lumbar puncture

CONTACTS AND LOCATIONS:
Overall Officials: Karl Alstadhaug, MD, PhD, Principal Investigator — Nordlandssykehuset HF; Francis Odeh, MD, PhD, Principal Investigator — Nordlandssykehuset HF
Locations (1):
- Departement of Neurology, NLSH HF, Bodø, Norway